CLINICAL TRIAL: NCT01750788
Title: Xarelto® on Prevention of Stroke and Non-central Nervous System Systemic Embolism in Patients With Non-valvular Atrial Fibrillation in Asia: A Non-interventional Study
Brief Title: Xarelto for Prevention of Stroke in Patients With Atrial Fibrillation in Asia
Acronym: XANAP
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16371; XA1205 (Other: Company internal)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation
Keywords: Stroke; Embolism; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Embolism | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Patients with non-valvular atrial fibrillation who are prescribed rivaroxaban under routine treatment conditions to prevent stroke or non-central nervous system systemic embolism. Decision regarding dose and duration of treatment made at the discretion of the attending investigator.

SUMMARY:
This is an international observational study in patients with non-valvular atrial fibrillation who are prescribed rivaroxaban under routine treatment conditions to prevent stroke or non-central nervous system systemic embolism.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 18 years of age with a diagnosis of non-valvular atrial fibrillation who start treatment with rivaroxaban to prevent stroke or non-CNS (Central Nervous System) systemic embolism, and who consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of non-valvular atrial fibrillation who start treatment with rivaroxaban to prevent stroke or non-CNS systemic embolism
Sampling Method: Probability Sample
Enrollment: 2297 (Actual)
Dates: Start 2013-01-13 (Actual); Primary Completion 2015-10-12 (Actual); Study Completion 2015-10-12 (Actual)

PRIMARY OUTCOMES:
Adjudicated major bleeding events | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Safety variables will be summarized using descriptive statistics based on adverse events collection | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
All cause mortality | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later

SECONDARY OUTCOMES:
Adjudicated symptomatic thromboembolic events | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Non-major bleeding, collected as SAEs or non-serious AEs and defined as all bleeding events that do not fall in the category of major bleedings | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Treatment satisfaction as per patient assessment of rivaroxaban treatment by the physician at the final visit | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Healthcare resource | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
  Number of healthcare professional visits and hospitalizations due to anticoagulation
Adverse events rates in the different AF risk factor categories | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Persistence with rivaroxaban treatment measured as percentage of patients on rivaroxaban treatment at 1 year after start of study treatment | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Reasons for switch of rivaroxaban treatment as per physician assessment during or at end of study | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later
Reasons for interruption of rivaroxaban treatment as per physician assessment during or at end of study | after 1 year or until 30 days after end of rivaroxaban therapy, whichever is later

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Many Locations, Hong Kong
- Many Locations, India
- Many Locations, Indonesia
- Many Locations, Malaysia
- Many Locations, Pakistan
- Many Locations, Philippines
- Many Locations, Singapore
- Many Locations, South Korea
- Many Locations, Taiwan
- Many Locations, Thailand
- Many Locations, Vietnam

REFERENCES:
- [Derived] Kirchhof P, Haas S, Amarenco P, Turpie AGG, Bach M, Lambelet M, Hess S, Camm AJ. Causes of death in patients with atrial fibrillation anticoagulated with rivaroxaban: a pooled analysis of XANTUS. Europace. 2024 Jul 2;26(7):euae183. doi: 10.1093/europace/euae183. PMID 38941511
- [Derived] Kirchhof P, Radaideh G, Kim YH, Lanas F, Haas S, Amarenco P, Turpie AGG, Bach M, Lambelet M, Hess S, Camm AJ; Global XANTUS program Investigators. Global Prospective Safety Analysis of Rivaroxaban. J Am Coll Cardiol. 2018 Jul 10;72(2):141-153. doi: 10.1016/j.jacc.2018.04.058. PMID 29976287